CLINICAL TRIAL: NCT07280897
Title: Implementation and Evaluation of SCIPI: A Multi-Site Pilot Randomized Controlled Trial to Improve Decision-Making and Quality of Life Among Patients With Localized Prostate Cancer
Brief Title: SCIPI Implementation and Evaluation: A Multi-site Proof-of-Concept Pilot Trial
Acronym: SCIPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Kansas Medical Center (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Lixin Song, Tenured Full Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00001556; E06709.1a (Other Grant/Funding Number: Department of Defense (DOD))
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either the SCIPI intervention or usual care. Randomization will be stratified by study site (KUMC, UCSD, UNC, UTHSA), and implemented in REDCap using permuted blocks with variable block sizes. Each participant remains in the assigned group for the duration of the study; there is no crossover.
Who Masked: Outcomes Assessor
Masking Description: Data collection staff are masked to group assignment; participants and providers are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCIPI (Experimental): Participants will receive SCIPI, a web-based supportive care program delivered through the Epic MyChart system, in addition to usual care.
  Interventions: Behavioral: SCIPI
- Usual Care (No Intervention): Participants will receive usual care provided at their study site.

INTERVENTIONS:
Behavioral: SCIPI — SCIPI (Support, Communication, and Information Program for Prostate Cancer - Interactive) is a web-based supportive care program delivered through the Epic MyChart system. The program provides tailored educational materials, skills training, and interactive tools to support informed treatment decision-making for patients with localized prostate cancer.
  Arms: SCIPI

SUMMARY:
This study will test a web-based supportive care program called the Support, Communication, and Information Program for Prostate Cancer - Interactive (SCIPI). SCIPI provides men with localized prostate cancer and their families with easy-to-understand information, tools to prepare for discussions with their doctors, and opportunities for social support. The purpose of this pilot study is to determine whether it is feasible to integrate SCIPI in prostate cancer clinical care via the electronic medical record and whether SCIPI may improve patients' confidence in making treatment decisions and their overall quality of life compared with usual care. The study will include patients who are newly diagnosed with prostate cancer. Participants will be randomly assigned to use SCIPI or to receive usual care, and information will be collected over time about their experiences, decision-making, and quality of life.

DETAILED DESCRIPTION:
This proof-of-concept pilot randomized clinical trial aims to test the feasibility and preliminary efficacy of SCIPI, a web-based supportive care intervention for patients with localized prostate cancer. The study will enroll 200 newly diagnosed patients across four NCI-designated cancer centers, with the option for family members to participate. After providing informed consent and completing the baseline assessment (T1), participants will be randomly assigned to either the SCIPI intervention or usual care. Data will be collected at 3 months (T2) and 6 months (T3) to evaluate decision satisfaction, quality of life, symptom burden, self-efficacy, and program usability.

ELIGIBILITY:
Inclusion Criteria:

Patients with localized prostate cancer:

* Age ≥ 18 years.
* Biopsy-confirmed diagnosis of localized prostate cancer (Gleason score ≤8, PSA < 30 ng/mL).
* Eligible for curative-intent treatment (e.g., surgery, radiation, or active surveillance).
* Able to read and understand English or Spanish.
* Access to the internet and the Epic MyChart patient portal at a participating study site (UTHSA, UNC, UCSD, or KUMC).
* Willing and able to provide informed consent.

Exclusion Criteria:

Patients:

* History of metastatic or recurrent prostate cancer.
* Diagnosis of another active malignancy (excluding non-melanoma skin cancer).
* Severe cognitive impairment or psychiatric illness that would interfere with participation.
* Inability to access the internet or the MyChart portal.
* Prior participation in other related digital health trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2029-09-29 (Estimated); Study Completion 2029-09-29 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Decision (SWD) | 3-month follow-up (T2) and 6-month follow-up (T3)
  SWD will be assessed using the 6-item Satisfaction with Decision (SWD) scale, which measures the extent to which participants feel informed, confident, and satisfied with their prostate cancer treatment decision. Scores range from 6 to 30, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Quality of Life (FACT-G) | Baseline (T1), 3-month follow-up (T2), 6-month follow-up (T3)
  Quality of life will be measured using Functional Assessment of Cancer Therapy - General (FACT-G). A 27-item validated questionnaire assessing physical, social/family, emotional, and functional well-being. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Song, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio School of Nursing, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with colleagues at all participating sites and with other researchers as requested and approved by the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be available for sharing after study completion and final data analysis. Summary results will be posted on ClinicalTrials.gov within one year after the study reaches its Primary Completion Date. Published data will be shared once the corresponding manuscript has been accepted and published in a peer-reviewed journal.